CLINICAL TRIAL: NCT00000904
Title: A Phase I Trial to Compare the Safety and Immunogenicity of the Live Recombinant Canarypox ALVAC-HIV Vaccines, vCP205, vCP1433, and vCP1452, in HIV-1 Uninfected Adult Volunteers
Brief Title: Safety and Effectiveness of Anti-HIV Vaccines in HIV-Negative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 034; AVEG 034A; 10583 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Viral Vaccines; HIV Antibodies; HIV Envelope Protein gp160; AIDS Vaccines; T-Lymphocytes, Cytotoxic; HIV Seronegativity; Antibody Formation; Risk-Taking; Avipoxvirus; Genetic Vectors; Immunization; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Risk-Taking

INTERVENTIONS:
Biological: ALVAC(2)120(B,MN)GNP (vCP1452)
Biological: gp160 MN/LAI-2
Biological: ALVAC(1)120(B,MN)GNP (vCP1433)
Biological: ALVAC-HIV MN120TMG (vCP205)
Biological: ALVAC-RG Rabies Glycoprotein (vCP65)

SUMMARY:
The purpose of this study is to find out whether three different anti-HIV vaccines are safe and whether they help prevent HIV infection. These vaccines are called vCP205, vCP1433, and vCP1452. Some patients also receive another anti-HIV vaccine, gp160. The vaccines are made up of small pieces of HIV, which help the body learn to recognize and destroy HIV. You cannot get HIV from these vaccines.

There are two different ways a vaccine can protect the body from infection. First, a vaccine may help the immune system make antibodies, which are proteins that recognize invading viruses or bacteria. Second, a vaccine may help the body make immune cells that destroy infected cells. The second type of vaccine is more powerful against HIV. In this study, doctors will see whether vCP205, vCP1433, vCP1452, and gp160 are good vaccines by seeing whether they help the body make immune cells.

DETAILED DESCRIPTION:
Previous studies in humans have shown that immunization with certain vaccine combinations (that is, ALVAC-HIV construct and an envelope subunit vaccine) can elicit CTL activity, antibody-dependent cellular toxicity (ADCC), neutralizing antibodies, and other antibody responses more often and at higher levels than either vaccine alone. This study examines improved vaccine candidates that can elicit broader, longer-lasting CTL activity in the majority of vaccine recipients.

Volunteers are randomized to one of four groups. Group I receives vCP205. Group II receives vCP1433. Group III receives vCP1452. Group IV receives an ALVAC rabies vaccine, as a control. Immunizations are administered at Months 0, 1, 3, and 6. At Months 3 and 6, patients in Groups I, II, and III also receive gp160 MN/LAI-2, the subunit boost vaccine. Group IV receives another placebo vaccine. Participants have regular clinic visits and blood is drawn to determine humoral and cellular immune responses to the vaccines. [AS PER AMENDMENT 10/23/98: A cell-mediated immunity substudy has been added at selected institutions following the fourth vaccination at 6 months; this study will assess the newer assays of CD8+ T cells and the kinetic response following immunization. The 6-month immunization may be rescheduled by up to 14 days to accommodate clinical, laboratory, or volunteer scheduling issues.] [AS PER AMENDMENT 6/17/99: Three study arms are added. Group V receives vCP1452 at Months 0,1,3, and 6. Group VI receives vCP205 at Months 0,1,3, and 6. Group VII receives placebo at Months 0,1,3, and 6. Patients in Groups V, VI, and VII do not receive the subunit boost, gp160 MN/LAI-2. Consenting volunteers enrolled in the three new groups at Johns Hopkins University undergo PET scanning as part of an ancillary study.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are 18-60 years old.
* Are HIV-negative and are in good health.
* Have a CD4 count of at least 400 cells/mm3.
* Test negative for hepatitis B.
* Agree to use effective methods of birth control for 1 month before and during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Are at high risk for being infected with HIV (risky sex behavior or injection drug use within 12 months prior to study entry).
* Have a serious medical condition, or if you have had chronic sickness, diseases of the immune system, or cancer that was not cured through surgery.
* Have a serious psychiatric condition or if you have been suicidal.
* Have a work commitment that would keep you from completing the study.
* Have syphilis or tuberculosis.
* Are allergic to eggs, neomycin, vaccines, or have ever had severe allergic reactions.
* Have taken certain medicines, including medicines that affect the immune system or experimental medicines.
* Have participated in another HIV vaccine trial.
* Have received any vaccines within 2 weeks of study entry.
* Have received a blood transfusion within 6 months prior to study entry.
* Are pregnant or breast-feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Study Completion 1999-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schwartz, Study Chair — Johns Hopkins Bloomberg School of Public Health; Clayton Harro, Study Chair — Johns Hopkins Bloomberg School of Public Health
Locations (6):
- United States (6):
  - UAB AVEG, Birmingham, Alabama
  - JHU AVEG, Baltimore, Maryland
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Fang ZY, Limbach K, Tartaglia J, Spearman P. A canarypox HIV vaccine candidate elicits efficient gag-env pseudovirion formation from human muscle cells. 36th Annual Meeting, Infectious Diseases Society of America. 1998 Nov 12-15 [Poster 710]
- [Background] Bures R, Gaitan A, Zhu T, Graziosi C, McGrath KM, Tartaglia J, Caudrelier P, El Habib R, Klein M, Lazzarin A, Stablein DM, Deers M, Corey L, Greenberg ML, Schwartz DH, Montefiori DC. Immunization with recombinant canarypox vectors expressing membrane-anchored glycoprotein 120 followed by glycoprotein 160 boosting fails to generate antibodies that neutralize R5 primary isolates of human immunodeficiency virus type 1. AIDS Res Hum Retroviruses. 2000 Dec 10;16(18):2019-35. doi: 10.1089/088922200750054756. PMID 11153085